CLINICAL TRIAL: NCT02693301
Title: Effects of an Intra-hospital Exercise Program for Children With Asthma and Respiratory Symptoms
Brief Title: Effects of an Exercise Program for Children With Asthma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Europea de Madrid (Other)
Responsible Party: Principal Investigator, Margarita Perez, Professor in Exercise Physiology, Universidad Europea de Madrid
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R-0031/14A
Record Dates: First submitted 2016-02-02; First posted 2016-02-26 (Estimated); Last update posted 2020-02-28 (Actual); Status verified 2020-02

CONDITIONS: Asthma
Keywords: Asthma; Respiratory symptoms; Exercise program; Functional capacity; Body composition
MeSH Terms: conditions — Asthma; Signs and Symptoms, Respiratory | interventions — Resistance Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Children who follow the recommendations of their pneumologist
- Experimental (Experimental): A two month intervention program 3 days/week will be carried out. The session will last ~60 minutes, and will consist of a combined training (aerobic training ~30 min, and strength ~30 min of 7 whole body exercises (3 sets x 10 repetitions).The load was gradually increased as the strength of each child improved, i.e., from 40% of five-repetition maximum (5RM) lifting ability at the start of the program to 60% of 5RM at the end of the program. All sessions were individually supervised by trained professionals.
  Interventions: Other: Exercise program

INTERVENTIONS:
Other: Exercise program
  Arms: Experimental

SUMMARY:
exercise program in the pulmonary function and cardiorespiratory fitness in children with asthma and respiratory symptoms

DETAILED DESCRIPTION:
This study aims to analyze the effects of an exercise program in the pulmonary function, cardiorespiratory fitness, diet quality index, physical activity, body composition, muscle function, agility, and psychological health in a group of children with asthma and respiratory symptoms

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with Asthma following the GEMA 2009 criteria (Spanish Guide for Asthma Management) at least 6 months prior to the study.
* Complete successfully both Cardiorespiratory and Functional Tests.

Exclusion Criteria:

* Diagnosed with other chronic respiratory disease or condition
* Diagnosed with any chronic disease including cardiovascular diseases.
* Reduced mobility
* Uncooperative
* Poor adherence to medication

Ages: 7 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 53 (Actual)
Dates: Start 2016-01; Primary Completion 2018-05 (Actual); Study Completion 2018-10 (Actual)

PRIMARY OUTCOMES:
Change in Pulmonary Function (Lung Function) | Baseline, 2 months, and 3 months
  Change from baseline to 2 months, and 3 months
Change in Cardiorespiratory Fitness | Baseline, 2 months, and 3 months
  Change from baseline to 2 months, and 3 months using Cardiorespiratory Test
Change in Muscle Strength | Baseline, 2 months, and 3 months
  Change from baseline to 2 months, and 3 months using one repetition maximum test
Change in Quality of life and anxiety status | Baseline, 2 months, and 3 months
  Change from baseline to 2 months, and 3 months using the Paediatric Asthma Quality of Life Questionnaire (PAQLQ) (Guyatt GH, 1997)
Change in anxiety | Baseline, 2 months, and 3 months
  Change from baseline to 2 months, and 3 months using STAIC (State-Trait Anxiety Inventory for Children)
Change in Body Mass Index (BMI) | Baseline, 2 months, and 3 months
  Change from baseline to 2 months, and 3 months using height and weight.
Change in Waist-to-Height index | Baseline, 2 months, and 3 months
  Change from baseline to 2 months, and 3 months using height and waist.
Change in anthropometric outcomes | Baseline, 2 months, and 3 months
  Change from baseline to 2 months, and 3 months using skinfolds, and circumferences.
Change in Body Composition | Baseline, 2 months, and 3 months
  Change from baseline to 2 months, and 3 months using Bioimpedance.
Changes in Physical Activity using questionnaires | Baseline, 2 months, and 3 months
  Change from baseline to 2 months, and 3 months using Physical Activity Questionnaire for Children (PAQ-C) and Adolescents (PAQ-A)
Change in Agility walking | Baseline, 2 months, and 3 months
  Change from baseline to 2 months, and 3 months using Test of Up and Go
Change in Agility stairs. | Baseline, 2 months, and 3 months
  Change from baseline to 2 months, and 3 months using Test of Up and Down Stairs (TUDS)

CONTACTS AND LOCATIONS:
Overall Officials: Margarita Perez Ruiz, MD, PhD, Principal Investigator — Universidad Europea de Madrid
Locations (1):
- Hospital Infantil Universitario Niño Jesus, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No